CLINICAL TRIAL: NCT03350035
Title: A Double-Blind Randomized, Placebo Controlled Study to Evaluate the Safety, Tolerability, Efficacy, and Pharmacokinetics of Intravenous Ganaxolone as Adjunctive Therapy to Treat Subjects With Status Epilepticus
Brief Title: Intravenous Ganaxolone as Adjunctive Therapy to Treat Subjects With Status Epilepticus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Marinus Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1042-SE-2001
Record Dates: First submitted 2017-11-17; First posted 2017-11-22 (Actual); Results first posted 2022-12-15 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Status Epilepticus; Convulsive Status EPILEPTICUS; Non Convulsive Status Epilepticus; Epilepsy
MeSH Terms: conditions — Status Epilepticus; Epilepsy

STUDY DESIGN:
Intervention Model Description: Double-blind study that will randomize subjects to ganaxolone or placebo in a 1:1 ratio as adjunctive therapy to their standard of care.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IV Ganaxolone active (Experimental): Ganaxolone IV loading dose with continuous infusion (maintenance dose) for 2-4 days followed by an 18-hour taper.
  Interventions: Drug: IV Ganaxolone active
- IV Placebo, non-active (Placebo Comparator): Placebo IV loading dose with continuous infusion (maintenance dose) for 2-4 days followed by an 18-hour taper.
  Interventions: Drug: IV Placebo, non-active

INTERVENTIONS:
Drug: IV Ganaxolone active — IV
  Arms: IV Ganaxolone active
Drug: IV Placebo, non-active — IV
  Arms: IV Placebo, non-active

SUMMARY:
This study will evaluate the effectiveness and safety of an investigational drug, IV ganaxolone, as adjunctive therapy to standard of care to treat subjects with status epilepticus.

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled study to evaluate the safety, tolerability, and efficacy of adjunctive IV ganaxolone in subjects with SE.

Study drug will be added to standard of care before IV anesthetic during the treatment of SE.

Subjects will be screened for inclusion/exclusion criteria prior to receiving study drug as adjunctive therapy by continuous IV. Subject's will be followed up for 3 weeks post-treatment.

Subjects who are known to be at risk for SE may be consented and/or assented prior to an SE event.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 12 years of age and older
* Clinical and/or electrographic seizures

Exclusion Criteria:

* Life expectancy of less than 24 hours
* Anoxic brain injury as primary cause of SE
* Recent (<24 hour) traumatic brain injury as the primary cause of SE
* Administered anesthesia for the treatment of SE

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2019-09-18 (Actual); Study Completion 2019-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maciej Gasior, MD, PhD, Study Director — Marinus Pharmaceuticals
Locations (8):
- United States (8):
  - Nemours/AI duPont Hospital for Children, Wilmington, Delaware
  - Nicklaus Children's Hospital, Miami, Florida
  - Grady Hospital, Atlanta, Georgia
  - Oschner Clinic Foundation, New Orleans, Louisiana
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Duke Medical Center, Durham, North Carolina
  - Allegheny General Hospital, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Vaitkevicius H, Ramsay RE, Swisher CB, Husain AM, Aimetti A, Gasior M. Intravenous ganaxolone for the treatment of refractory status epilepticus: Results from an open-label, dose-finding, phase 2 trial. Epilepsia. 2022 Sep;63(9):2381-2391. doi: 10.1111/epi.17343. Epub 2022 Jul 10. PMID 35748707

RESULTS

PARTICIPANT FLOW:
Groups:
- Low - GNX: 500 mg/day
- Medium - GNX: 650 mg/day
- High - GNX: 713 mg/day
Period: Overall Study
Arm/Group | Low - GNX | Medium - GNX | High - GNX
Started | 5 | 4 | 8
Completed | 3 | 4 | 7
Not Completed | 2 | 0 | 1
Not completed — Lack of Efficacy | 2 | 0 | 0
Not completed — Subject discharged to hospice | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Low - GNX | Medium - GNX | High - GNX | Total
Number analyzed (Participants) | 5 | 4 | 8 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.8 (25.35) | 62.0 (18.96) | 53.8 (17.04) | 56.9 (19.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 2 | 9
  Male | 0 | 2 | 6 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 4 | 6 | 15
  Unknown or Not Reported | 0 | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 2 | 5
  White | 3 | 2 | 4 | 9
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Did Not Require an IV Anesthetic Drug for SE Treatment
Description: Number of participants who did not require an intravenous (IV) Anesthetic Drug (a third-line Treatment) for Status Epilepticus (SE) within the first 24 hours after Study Drug Initiation.
Time Frame: 24 hours post study drug initiation
Population: Safety Population: included all participants who received at least one dose of IV ganaxolone (GNX).
Measure: Count of Participants; unit: Participants
Arm/Group | Low - GNX | Medium - GNX | High - GNX
Number analyzed (Participants) | 5 | 4 | 8
Participants | 5 | 4 | 8

2. Secondary Outcome: Time to Cessation of SE
Description: Summary of Time to SE Cessation
Time Frame: Time to SE Cessation, assessed up to 24 hours
Population: Safety Population. Only participants were included if seizure was confirmed.
Measure: Median (Full Range); unit: Minutes
Arm/Group | Low - GNX | Medium - GNX | High - GNX
Number analyzed (Participants) | 5 | 4 | 7
Minutes | 5.000 [2.45 to 6.05] | 5.580 [4.18 to 22.25] | 10.16 [1.34 to 241.00]

3. Secondary Outcome: Number of Participants Who Required No Escalation of Treatment for Ongoing or Recurrent SE
Description: Number of participants who Required No Escalation of Treatment for Ongoing or Recurrent SE
Time Frame: Drug initiation through follow-up period, up to approximately 4 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Low - GNX | Medium - GNX | High - GNX
Number analyzed (Participants) | 5 | 4 | 8
Participants | 3 | 3 | 8

4. Secondary Outcome: Number of Participants With No SE Recurrence Per Principal Investigator
Description: Number of participants with No SE Recurrence per Principal Investigator within 24hrs of starting treatment, during treatment period (excluding taper), during taper, during 24-hr follow-up period, and during follow-up period.
Time Frame: Baseline (within 24hrs of treatment) through follow up period, up to approximately 4 weeks.
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Low - GNX | Medium - GNX | High - GNX
Number analyzed (Participants) | 5 | 4 | 8
Participants
  Within 24hrs of starting treatment | 5 | 4 | 7
  During treatment period (excluding taper) | 3 | 4 | 7
  During taper | 3 | 2 | 7
  During 24-hr follow-up period | 3 | 3 | 8
  During follow-up period | 1 | 3 | 7

5. Secondary Outcome: Seizure Burden
Description: Seizure Burden (%) Baseline and Percentage Change from Baseline by Time Point
Time Frame: Baseline (Pre-dose) to <-24hrs (Post Dose)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Percentage change from baseline
Arm/Group | Low - GNX | Medium - GNX | High - GNX
Number analyzed (Participants) | 5 | 4 | 8
Percentage change from baseline
  Change from Baseline at 0 to <- 1 Hour Post-Dose: number analyzed (Participants) | 4 | 4 | 8
  Change from Baseline at 0 to <- 1 Hour Post-Dose | -94.80 (8.458) | -74.63 (25.247) | -84.01 (18.862)
  Change from Baseline at 0 to <- 4 Hour Post-Dose: number analyzed (Participants) | 4 | 4 | 8
  Change from Baseline at 0 to <- 4 Hour Post-Dose | -98.59 (2.092) | -71.75 (33.498) | -87.99 (21.439)
  Change from Baseline at >4 to <- 8 Hours Post-Dose: number analyzed (Participants) | 4 | 4 | 8
  Change from Baseline at >4 to <- 8 Hours Post-Dose | -77.53 (17.950) | -59.80 (48.352) | -96.58 (6.772)
  Change from Baseline at >8 to <- 16 Hours Post-Dose: number analyzed (Participants) | 4 | 4 | 8
  Change from Baseline at >8 to <- 16 Hours Post-Dose | -47.98 (38.063) | -53.29 (44.490) | -93.75 (13.306)
  Change from Baseline at >16 to <- 24 Hours Post-Dose: number analyzed (Participants) | 4 | 4 | 8
  Change from Baseline at >16 to <- 24 Hours Post-Dose | -99.53 (0.935) | -48.25 (45.475) | -81.16 (47.368)
  Change from Baseline at 0 to <- 24 Hours Post-Dose: number analyzed (Participants) | 4 | 4 | 8
  Change from Baseline at 0 to <- 24 Hours Post-Dose | -78.64 (15.286) | -56.10 (42.183) | -89.06 (20.039)

ADVERSE EVENTS:
Time Frame: Baseline (within 24hrs of treatment) through follow up period, up to approximately 4 weeks
Arm/Group | Low - GNX | Medium - GNX | High - GNX
All-Cause Mortality (participants affected / at risk) | 2/5 | 0/4 | 1/8
Serious Adverse Events (participants affected / at risk) | 2/5 | 2/4 | 2/8
Other Adverse Events (participants affected / at risk) | 5/5 | 3/4 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low - GNX (N=5) | Medium - GNX (N=4) | High - GNX (N=8)
Sedation (Nervous system disorders) | 0 | 1 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Endotracheal intubation (Surgical and medical procedures) | 1 | 0 | 0
Withdrawal of life support (Surgical and medical procedures) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Low - GNX (N=5) | Medium - GNX (N=4) | High - GNX (N=8)
Somnolence (Nervous system disorders) | 1 | 1 | 3
Sedation (Nervous system disorders) | 0 | 1 | 1
Pain (General disorders) | 1 | 1 | 0
Hypotension (Vascular disorders) | 2 | 0 | 2
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypercaprnia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Pneumonia (Infections and infestations) | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 1

LIMITATIONS AND CAVEATS:
2 deaths during the follow-up were extracted from the SAE reconciliation database.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-08-07): https://cdn.clinicaltrials.gov/large-docs/35/NCT03350035/Prot_002.pdf
  • Statistical Analysis Plan (2020-05-04): https://cdn.clinicaltrials.gov/large-docs/35/NCT03350035/SAP_003.pdf